CLINICAL TRIAL: NCT06870695
Title: Safety and Efficiency of Electrocautery De-Epithelization in Mammoplasty
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Elghazaly, Lecturer of Plastic and Reconstructive Surgery, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1061/1/25
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Safety; Efficiency; Electrocautery; De-Epithelization; Mammoplasty
MeSH Terms: interventions — Electrocoagulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electrocautery group: Patients undergoing standard surgical de-epithelization with electrocautery.
  Interventions: Procedure: Electrocautery
- Control group: Patients undergoing standard surgical de-epithelization using surgical blade by scalpel.
  Interventions: Procedure: Surgical blade by scalpel

INTERVENTIONS:
Procedure: Electrocautery — Patients undergoing standard surgical de-epithelization with electrocautery.
  Groups: Electrocautery group
Procedure: Surgical blade by scalpel — Patients undergoing standard surgical de-epithelization using surgical blade by scalpel.
  Groups: Control group

SUMMARY:
The aim of this study is to evaluate safety and efficiency of electrocautery de-epithelization in mammoplasty.

DETAILED DESCRIPTION:
Mammoplasty is the fifth most commonly performed by plastic surgeons worldwide to improve symptomatology resulting from macromastia.

One of the key stages in a breast reduction or augmentation surgery is the de-epithelization process. De-epithelialization is the first stage of reduction mammoplasty in techniques that use dermal, dermo-glandular pedicles. Traditional methods of de-epithelization include manual dissection or mechanical scraping as time-consuming and demanding by most surgeons, especially when the breasts are large and when there is no assistant available.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients undergoing mammoplasty.

Exclusion Criteria:

* Patients with active infections or open wounds at the surgical site.
* Individuals with known hypersensitivity or adverse reactions to electrocautery.
* Pregnant or lactating women.
* Patients with uncontrolled diabetes or coagulation disorders.
* History of psychiatric illness.
* Patients undergoing secondary or repeat breast reduction procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing mammoplasty
Study Population: This retrospective study was conducted on 100 females patients aged 18 years or older who were scheduled to undergo mammoplasty at Tanta University Hospitals, Egypt between July 2024 and February 2025
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperatively
  Operative time (time taken from skin incision to completion of skin closure). Operative time will be measured for each breast

SECONDARY OUTCOMES:
Degree of pain | 3 days after surgery
  Degree of pain will be measured using a standard 10-point visual analog pain scale (VAS). The women verbally reported a pain rating for each breast first in the recovery room (within 4 hours of surgical stop) and again at the first follow-up visit (1 to 3 days after surgery).
De-epithelization time | Intraoperatively
  De-epithelization time will be recorded.
Time to achieve hemostasis | Intraoperatively
  The time to achieve hemostasis will be assessed.
Duration of drain placement | Intraoperatively
  Duration of drain placement will be recorded.
Blood loss | Intraoperatively
  Blood loss will be assessed by weighing the swabs that will be used during the pedicle de-epithelialization process.
Wound healing time | 6 weeks after surgery
  Wound healing time will be recorded.
Incidence of adverse events | 6 weeks after surgery
  The incidence of adverse events such as flap necrosis, hematoma, seroma, and surgical site infection will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: The data will be available upon a reasonable request from the corresponding author.
Access Criteria: After the end of study for one year.